CLINICAL TRIAL: NCT06698822
Title: A Phase 2 Trial to Assess Safety and Efficacy of Tofacitinib 2% Cream in the Treatment of Cutaneous T-cell Lymphoma (CTCL), Stages IA, IB, and IIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0747; NCI-2024-09674 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tofacitinib 2% (Experimental): Participants will apply a thin layer of tofacitinib 2% cream 2 times a day on up to 5 treatment-eligible skin lesions.
  Interventions: Drug: tofacitinib 2% cream

INTERVENTIONS:
Drug: tofacitinib 2% cream — Given topical

SUMMARY:
To study the safety and effectiveness of tofacitinib 2% cream in treating early-stage CTCL.

DETAILED DESCRIPTION:
Primary Objectives

* To assess the safety of tofacitinib 2% cream in the treatment of early stage CTCL (stage IA, IB, or IIA)
* To assess the overall response rate (ORR) of target lesions at Week 12 based upon Modified Composite Assessment of Index Lesion Severity (mCAILS)

Secondary Objectives

* To assess the overall response rate (ORR) of target lesions at Week 12 based upon mSWAT composite score
* To assess response by mCAILS at weeks 20, 28, 36, 44, and 52 for participants that choose to extend treatment
* To assess the time to overall response by mCAILS score
* To assess the duration of overall response by mCAILS score
* To assess pruritus using the visual analog scale at baseline, 4 weeks, 8 weeks, and 12 weeks
* To assess health-related quality of life using the Skindex-29 instrument at baseline, 4 weeks, 8 weeks, and 12 weeks To characterize the JAK/STAT biomarker profile of tumors and characterize the mutational landscape in tumors before and after therapy

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at screening visit. Because limited dosing and adverse event data are currently available on the use of tofacitinib in participants <18 years of age, children are excluded from this study.

  * Have a clinical diagnosis of cutaneous T-cell lymphoma (CTCL) stage IA, IB, or IIA including documentation of a skin biopsy with histological findings consistent with CTCL.
  * For stage IIA, only participants with a classification of N0 (no clinically abnormal peripheral lymph nodes) or N1 (clinically abnormal lymph node(s) histopathology Dutch grade 1 or NCI LN0-2) can be enrolled.
  * Participants must be B0 (absence of significant blood involvement: .5% of peripheral blood lymphocytes of <250/mcL are atypical.
  * Have at least 2 distinct lesions that have either failed or recurred despite treatment with 1 previous standard therapy.
  * ECOG performance status ≤ 2 (Karnofsky .60%)
  * Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
  * The effects of tofacitinib on the developing human fetus are unknown. Available data with tofacitinib in its oral formulation in pregnant women are insufficient to establish a drug associated risk of major birth defects, miscarriage or adverse maternal or fetal outcomes. Therefore, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following:

    1. Postmenopausal (no menses in greater than or equal to 12 consecutive months)
    2. History of hysterectomy or bilateral salpingo-oophorectomy
    3. Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy)
    4. History of bilateral tubal ligation or another surgical sterilization procedure
  * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of tofacitinib administration.

    * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tofacitinib

  * Skin infection and/or skin ulceration at screening and baseline visit
  * Any subject with a diagnosis of active malignancy or a cancer requiring treatment of expected to require treatment during the course of the trial (not including basal cell carcinoma, squamous cell carcinoma of the skin, malignant melanoma in situ, or cervical carcinoma in situ)
  * Any uncontrolled or serious underlying disease or medical or surgical condition that may interfere with interpretation of the trial results and/or place the subject at significant risk according to investigator discretion including but not limited to severe cardiac, psychiatric, hematologic, and thyroid conditions
  * History of Stage IIB or greater CTCL, or stage IIA CTCL with history of stage N2 (Dutch Grade 2 or NCI LN3 or greater), or with >5% circulating Sezary cells
  * History of aggressive CD8+ CTCL disease
  * Having received one of the following treatments within the specified timeframes (calculated from baseline visit):

    * In the past 12 weeks: Total Skin Electron Beam Therapy (TSEBT)
    * In the past 8 weeks: topical imiquimod
    * In the past 4 weeks: topical corticosteroids, topical chemotherapy, topical retinoids, local radiation therapy, UVB therapy, PUVA, photopheresis, systemic retinoids, systemic corticosteroids, interferon inducers, systemic chemotherapeutic agents
  * Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia
  * Participants who are receiving any other investigational agents
  * Participants with uncontrolled intercurrent illness
  * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
  * Participants with psychiatric illness/social situations that would limit compliance with study requirements
  * Pregnant women are excluded from this study because the effects of tofacitinib on the developing human fetus are unknown. As there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with tofacitinib, breastfeeding should be discontinued if the mother is treated with tofacitinib. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AE's) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Julia Dai, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org